CLINICAL TRIAL: NCT05376072
Title: Efficacy of Electromyographic Biofeedback in Muscle Recovery After Meniscectomy in Soccer Players
Brief Title: Electromyographic Biofeedback Muscle Recovery Meniscectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Norway University of Applied Sciences (Other)
Collaborators: University of Malaga (Other)
Responsible Party: Principal Investigator, Coral Falco, Principal Investigator, Western Norway University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Biofeedback_UMA-WNUAS_2022
Record Dates: First submitted 2022-05-02; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Feedback, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental data (Experimental)
  Interventions: Other: Electromyographic Biofeedback

INTERVENTIONS:
Other: Electromyographic Biofeedback — The players performed 10 work sessions with EMG-BF. Each session was divided into three phases: (a) three trials without receiving feedback, (b) between six and ten trials with feedback of electromyographic activity, (c) three trials without feedback. In each trial, isometric contractions of the vastus lateralis were performed.
  During maximum effort isometric contraction, the software associated with the ProComp Infiniti biofeedback unit collects the amplitude, the mean and maximum electromyographic signal, and also the contraction and tightening times. The contrac-tion time comprises the interval between the start of the contraction and achievement of the desired muscle tension. The tightening time is the period in which the tension voluntarily reached is maintained. For this study, the maximum and mean elec-tromyographic activity values were considered, calculated during the muscle tension time and maintained during each trial.

SUMMARY:
Electromyographic biofeedback (EMG-BF) is a therapeutic technique that has been used success-fully in rehabilitation of injuries. Although it has been applied in athletes, its use in this field is not very widespread. The objective of this study is to analyze its effectiveness in the recovery of electromyographic activity of the quadriceps after meniscectomy, evaluated through isometric contraction of the vastus lateralis. The sample comprised ten professional footballers in the Spanish League (2nd Division A) who had previously suffered a meniscus injury in their knee and had undergone a meniscectomy. The intervention consisted of EMG-BF treatment lasting between 6 and 10 sessions. The electromyographic signal was recorded using a Thought Tech-nology ProComp Infiniti 8-channel biofeedback unit with a sampling rate of 2048 sam-ples/seconds. For each session a within-subject ABA design of 6 or 10 trials per session was used, with three pre- and three post-measures, which determined the gain for each session.

ELIGIBILITY:
Inclusion Criteria:

* Partial meniscus tear
* Meniscectomy

Exclusion Criteria:

* Having an injury other than a partial meniscus tear

Ages: 24 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in muscle tension level | Each participant performed a total of 10 session during 5 weeks
  Using electrommiographic biofeedback device, the increase in muscle tension after isometric contraction was observed.
  Each player performed 10 work sessions (2 sessions per week) with EMG-BF. Each session was divided into three phases: (a) three trials without receiving feedback, (b) between six and ten trials with feedback of electromyographic activity, (c) three trials without feedback.
  In each trial, isometric contractions of the vastus lateralis were performed. For all sessions, each isometric contraction lasted six seconds and the participants rested for two minutes between trials to recover their contraction capacity. The sampling rate was 2048 samples per second.

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio Hernández Mendo, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Undecided